CLINICAL TRIAL: NCT06522542
Title: Retrospective Study on Anti-cancer Therapy for Gastric Cancer Patients Complicated With Bleeding
Brief Title: Gastric Cancer Complicated With Bleeding
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Yanhong Yao, Department of Medical Oncology and Radiation Sickness, Peking University Third Hospital
Other Study IDs: IRB00006761-M2023544
Record Dates: First submitted 2024-07-19; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: Gastirc cancer with bleeding at first diagnosis
  Interventions: Drug: systematic therapy
- Control group: Gastirc cancer without bleeding at first diagnosis
  Interventions: Drug: systematic therapy

INTERVENTIONS:
Drug: systematic therapy — All patients received systematic therapy including chemotherapy, targeted therapy or immune checkpoint inhibitor. We aims to investigate the impact of bleeding on the survival and treatment-related adverse events (TRAEs) of gastric cancer patients.
  Other Names: chemotherapy, targeted therapy or immune checkpoint inhibitor

SUMMARY:
To investigate the impact of bleeding on the survival and treatment-related adverse events (TRAEs) of gastric cancer patients.

DETAILED DESCRIPTION:
We will retrospectively enroll patients diagnosed with advanced or metastatic gastric cancer at the Department of Medical Oncology and Radiation Sickness of Peking University Third Hospital. The retrospective study aims to investigate the impact of bleeding on treatment-related adverse events (TRAEs) for gastric cancer patients receiving systematic anticancer treatment, assess the influence of bleeding on the survival of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years;
2. A histologically confirmed diagnosis of advanced or metastatic gastric cancer;
3. The initial anticancer treatment was systematic therapy, including chemotherapy, targeted therapy or immune checkpoint inhibitor (ICI);
4. No history of gastrectomy before systematic therapy.

Exclusion Criteria:

1. Incompletable clinical data;
2. Siewert I type esophagus cancer.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Advanced or metastatic gastric cancer at the Department of Medical Oncology and Radiation Sickness of Peking University Third Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | from date of the first cycle of systematic therapy to death from any cause，assessed up to 120 months
  OS was defined as the time from the first cycle of systematic therapy to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Yao, Principal Investigator — Department of Medical Oncology and Radiation Sickness, Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Yes
The datasets analyzed during the study are available on reasonable request.
Supporting Information: CSR
Time Frame: After the trial is completed
Access Criteria: Used for scientific research

REFERENCES:
- [Derived] Yao Y, Liu Z, Zhang H, Shi X, Huang F, Zhang Y, Chen L, Shi Y, Cao B. Feasibility of systemic therapy in unresectable gastric/gastroesophageal junction cancer with overt bleeding. Asia Pac J Oncol Nurs. 2025 Jul 7;12:100750. doi: 10.1016/j.apjon.2025.100750. eCollection 2025 Dec. PMID 40747247

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT06522542/Prot_SAP_000.pdf